CLINICAL TRIAL: NCT06558539
Title: Study on the Efficacy of Wearable Transcutaneous Tibial Nerve Stimulation for Persistent Overactive Bladder Symptoms Post Benign Prostatic Hyperplasia Surgery
Brief Title: Tibial Nerve Stimulation for Post-BPH Overactive Bladder
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qing Yuan (Other)
Responsible Party: Sponsor-Investigator, Qing Yuan, Associate Chief Physician of Urology, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTNS2024
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Persistent Overactive Bladder Symptoms Post Benign Prostatic Hyperplasia Surgery
MeSH Terms: interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combination Therapy (Experimental): Approximately 30 participants are expected to be enrolled, and they will receive a combination of standard medication and TTNS therapy for 12 weeks.
  Interventions: Combination Product: Combination Therapy
- TTNS (Experimental): Approximately 30 participants are expected to be enrolled, and they will receive TTNS therapy for 12 weeks.
  Interventions: Device: Transcutaneous Tibial Nerve Stimulation(TTNS)
- Standard Medication Therapy (Active Comparator): Approximately 30 participants are expected to be enrolled, and they will receive standard medication and TTNS therapy for 12 weeks.
  Interventions: Drug: Standard Medication Therapy

INTERVENTIONS:
Device: Transcutaneous Tibial Nerve Stimulation(TTNS) — Participants in this group will discontinue all relevant medications (e.g., β3-adrenergic agonists, non-selective β-adrenergic agonists, or anticholinergic drugs) at least 14 days before signing the informed consent and will not use these medications during the study period. They will receive treatment solely with wearable transcutaneous tibial nerve stimulation.
  Arms: TTNS
Combination Product: Combination Therapy — Participants in this group will continue their prescribed medication regimen, which may include β3-adrenergic agonists, non-selective β-adrenergic agonists, or anticholinergic drugs, with dosages and administration unchanged throughout the study. In addition to the standard medication therapy, participants will receive wearable transcutaneous tibial nerve stimulation using a wearable device
  Arms: Combination Therapy
Drug: Standard Medication Therapy — Participants in this group will maintain their usual medication regimen, which may include β3-adrenergic agonists, non-selective β-adrenergic agonists, or anticholinergic drugs, with dosages and administration remaining consistent throughout the study. No additional interventions will be provided.
  Arms: Standard Medication Therapy

SUMMARY:
A single-center, randomized, parallel-controlled design. Approximately 90 cases of persistent overactive bladder symptoms post benign prostatic hyperplasia surgery are expected to be enrolled. The study participants will be randomly assigned to three groups, with 30 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with overactive bladder before benign prostatic hyperplasia 2.Overactive bladder still exists 1 month after the operation of benign prostatic hyperplasia; 3.50 ≤ age ≤80 , male 4.72-hour urination diary showed an average of ≥8 urination times every 24 hours at baseline

Exclusion Criteria:

-

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Average Daily Urination Frequency Compared to Baseline | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the change in average daily urination frequency compared to baseline will be calculated using the participants' 72-hour voiding diaries

SECONDARY OUTCOMES:
Average Urinary Urgency Score | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the average urinary urgency score will be calculated using the participants' 72-hour voiding diaries
Average Daily Nocturia Frequency Compared to Baseline | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the change in average daily nocturia frequency compared to baseline will be calculated using the participants' 72-hour voiding diaries
Average Voided Volume per Urination Compared to Baseline | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the change in average voided volume per urination compared to baseline will be calculated using the participants' 72-hour voiding diaries
Average Daily Incontinence Episodes | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the average daily incontinence episodes will be calculated using the participants' 72-hour voiding diaries
OABSS Compared to Baseline | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the change in Overactive Bladder Symptom Score (OABSS) compared to baseline will be calculated.
PPBC-S Compared to Baseline | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the change in Patient Perception of Bladder C Scale (PPBC-S) compared to baseline will be calculated.
AUA-SI-QOL Compared to Baseline | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the change in American Urological Association- Symptom Index-Quality of life (AUA-SI-QOL) compared to baseline will be calculated.
SAS Compared to Baseline | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, the change in Self-Rating Anxiety Scale (SAS) compared to baseline will be calculated.
Participant Satisfaction | treatment during 12 weeks : assessments at weeks 4, 8, and 12.
  At the end of Weeks 4, 8, and 12, participant satisfaction will be assessed using a participant satisfaction questionnaire
Potential Adverse Events Related by TTNS | Entire Study
  During the study, information on potential adverse events related to TTNS will be recorded, including pain and infection at the stimulation site, tibial nerve injury (such as motor dysfunction, neuralgia, etc.), urinary system complications (such as urinary retention), and other adverse events that the investigator deems potentially related to TTNS."